CLINICAL TRIAL: NCT04690335
Title: A Randomised, Phase 2a, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Prophylactic Efficacy of MV-012-968 Against Respiratory Syncytial Virus (RSV) Infection in the Virus Challenge Model.
Brief Title: Human Challenge Study to Evaluate the Efficacy of MV-012-968 Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meissa Vaccines, Inc. (Industry)
Collaborators: Hvivo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MV-004; 2020-002848-22 (EudraCT Number)
Record Dates: First submitted 2020-12-28; First posted 2020-12-30 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: RSV Infection
Keywords: RSV; vaccine; live attenuated; intranasal; challenge; Phase 2; safety; efficacy
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MV-012-968 (Experimental): Dose: 1 x10^6 Plaque Forming Unit (PFU), given intranasally, followed approximately 28 days later by inoculation with RSV-A (Memphis 37b).
  Interventions: Biological: MV-012-968
- Placebo (Placebo Comparator): Sodium Chloride 0.9% w/v intravenous infusion B.P (Normal Saline) matched to reference article product, given intranasally.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MV-012-968 — MV-012-968 is a recombinant, live attenuated RSV vaccine.
  Arms: MV-012-968
Other: Placebo — Saline solution
  Arms: Placebo

SUMMARY:
The purpose of this research study is to evaluate whether the investigational, live attenuated, intranasally delivered vaccine MV-012-968 ('study vaccine') may have prophylactic efficacy against symptomatic RSV infection when administered to adults 18-45 years of age in the Human Viral Challenge model.

ELIGIBILITY:
Key Inclusion Criteria:

1. An informed consent document signed and dated by the participant and the Investigator.
2. Aged between 18 and 45 years old on the day of signing the consent form.
3. In good general health with no history, or current evidence, of clinically significant medical conditions (including respiratory, cardiac and immunodeficiency), and no clinically significant test abnormalities that will interfere with participant safety, as defined by medical history, physical examination (including vital signs), electrocardiogram (ECG), and routine laboratory tests as determined by the Investigator.
4. A documented medical history prior to enrolment.
5. Females of child bearing potential must have a negative pregnancy test prior to enrollment.
6. Females and Males must agree to adhere to the highly effective contraceptive requirements of the study from 2 weeks prior to the first study visit until 90 days after the date of study vaccination.
7. Sero-suitable to the challenge virus, as defined in the study Analytical Plan.

Exclusion Criteria:

1. History of symptoms or signs suggestive of upper or lower respiratory tract infection within 4 weeks prior to the first study visit
2. Rhinitis which is clinically active
3. History of moderate to severe rhinitis
4. Acute sinusitis during Screening
5. Use of corticosteroid in respiratory tract (e.g. nasal or inhaled steroid) in the 30 days leading up to study vaccination
6. Females who are breastfeeding or have been pregnant within 6 months prior to the study
7. Participants who have smoked ≥ 10 pack years at any time [10 pack years is equivalent to one pack of 20 cigarettes a day for 10 years])
8. Positive human immunodeficiency virus (HIV), active hepatitis A (HAV), B (HBV), or C (HCV) test
9. Those employed or immediate relatives of those employed at hVIVO or the Sponsor
10. Participants may not live or work in direct close contact with, or live with anyone whose work brings them into direct close contact with, children under 2 years of age
11. Any other finding that, in the opinion of the Investigator, deems the participant unsuitable for the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Frequency of symptomatic RSV infection, as defined as the occurrence of both: | 10 days (days 2 to 12)
  * At least 1 quantifiable plaque assay sample in nasal wash specimens and
  * Symptoms meeting either: (i) a symptom of any grade from 2 different symptom categories from the participant Symptom Diary Card [SDC] (Upper Respiratory, Lower Respiratory, Systemic) or (ii) at least 1 Grade 2 upper or lower respiratory symptom from the participant SDC

SECONDARY OUTCOMES:
Frequency of symptomatic RSV infection, as defined as occurrence of both: | 10 days (days 2 to 12)
  * Two Quantifiable RT-qPCR samples on 2 consecutive days (i.e. at least 1 on each of 2 consecutive days) in nasal wash specimens and
  * Symptoms meeting either: (i) a symptom of any grade from 2 different symptom categories from the SDC (Upper Respiratory, Lower Respiratory, Systemic) or (ii) at least 1 Grade 2 upper or lower respiratory symptom from the participant SDC
Frequency of RSV infection, as defined as the occurrence of 2 quantifiable RT-qPCR samples on 2 consecutive days (i.e. at least 1 on each of 2 consecutive days) in nasal wash specimens | 10 days (Day 2 to 12)
Frequency of RSV infection, as defined as the occurrence of at least 1 quantifiable plaque assay sample in nasal wash specimens | 10 days (Day 2 to 12)
Mean daily total symptom score using the SDC | 10 days (Day 2 to 12)
Mean daily weight of nasal (mucus) discharge | 10 days (Day 2 to 12)
RSV load Area Under the Curve (AUC), as measured by RT-qPCR analysis of nasal wash specimens | 10 days (Day 2 to 12)
Peak RSV load, as measured by RT-qPCR of nasal wash specimens | 10 days (Day 2 to 12)
Frequency of solicited adverse events (AEs) as reported in the Subject Vaccination Diary Card, categorized by severity. Solicited AEs are predefined AEs that may occur after study vaccine administration. | Time Frame: 7 days (Day -28 to -21)
Frequency of unsolicited AEs after study vaccination, categorized by severity and by study vaccine relatedness. | 28 days (Day -28 to 0)
  Unsolicited AEs are any untoward medical occurrences in a participant administered the study vaccine, regardless of causal relationship to the study vaccine. Unsolicited AEs can include unfavorable and unintended signs (including abnormal laboratory findings), symptoms, or diseases temporally associated with the use of the study vaccine.
Frequency of unsolicited AEs after RSV-A challenge, categorized by severity and by study vaccine relatedness. | 29 days (Day 0 to 28)
Frequency of serious AEs (SAEs) after study vaccination, categorized by study vaccine relatedness. | 180 days (Day -28 to 152)
  SAEs are AEs, whether considered causally related to the study vaccine or not, that threaten life or result in any of the following: death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or congenital anomaly/birth defect.
Frequency of medically attended AEs (MAEs) after study vaccination, categorized by study vaccine relatedness. | 180 days (Day -28 to 152)
  MAEs are AEs, whether considered causally related to the study vaccine or not, with unscheduled medically attended visits, such as urgent care visits, acute primary care visits, emergency department visits, or other previously unplanned visits to a medical provider. Scheduled medical visits such as routine physicals, wellness checks, 'checkups', and vaccinations, are not considered MAEs

CONTACTS AND LOCATIONS:
Overall Officials: Mariya Kalinova, MD, Principal Investigator — hVIVO Services Ltd; Oliver Medzihradsky, MD MPH MS, Study Director — Meissa Vaccines, Inc.
Locations (1):
- hVIVO Services Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No